CLINICAL TRIAL: NCT00202007
Title: A Multi-Center, Randomized, Double-Blind Study, Comparing With Risperidone, to Evaluate the Efficacy and Safety of Aripiprazole in the Treatment of Patients With Schizophrenia
Brief Title: Efficacy and Safety Study of Aripiprazole to Treat Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Collaborators: Zhejiang Otsuka Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBRI0002
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2005-09

CONDITIONS: Schizophrenia
Keywords: Aripiprazole; Schizophrenia; Clinical trial; Risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Risperidone

INTERVENTIONS:
Drug: Aripiprazole tablet, 5-30mg/day, oral, 6 weeks
Drug: Risperidone tablet, 1-6mg/day, oral, 6 weeks

SUMMARY:
This study design is subject to relevant SFDA regulations about clinical trials. Patients will be screened for inclusion into the study at the initial visit(240 patients to be recruited) and then undergo a minimum of 3-7 day's placebo washout period(placebo wash out is to eliminate the effect of prior antipsychotic medication with tablets without any active ingredients)(patients without prior antipsychotic medication are exempt from the washout phase). After screening and washout period, eligible patients will be randomly assigned to the two treatment group, Aripiprazole or Risperidone, for 6 week's treatment. Patients will be hospitalized for the entire duration of the study. Patients' condition will be assessed weekly.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for screening

1. Schizophrenia or Acute schizophrenia-like psychotic disorder(ICD 10)
2. PANSS total of no less than 60
3. Age: 18-65; male or female
4. Informed consent from the legal guardians of the patients Inclusion criteria after washout

1.PANSS total of no less than 60 2.3-7days washout with placebo is required after discontinuation of other oral antipsychotics; No washout is needed for patients who had never taken any antipsychotics before; In cases that patients's condition is deemed clinically deteriorating and immediate treatment is needed, patients with less than 3 days' placebo washout could be randomized after notifying the sponsor 3.No serious function impairment in heart, liver or kidney.

-

Exclusion Criteria:

For screening

1. Tendency or history of suicide
2. Patients with extreme agitation, violent attacking behavior towards people and those who can hardly comply with treatment
3. Diagnosis of other mental diseases besides Schizophrenia
4. Diabetes or other serious unstable diseases or the following neurological diseases, migraine, epilepsy, Parkinson's disease, Alzheimer's disease, multiple sclerosis, stroke and TIA etc
5. Patients who take Fluoxetine in the past 1-month before screening
6. Patients who had participated any other clinical trial in the past 1-month before screening
7. History of alcohol or drug abuse or dependence
8. Pregnancy or breast-feeding
9. Patients who have had gastrointestinal operations that could affect drug absorption.
10. Allergy to Risperidone or Aripiprazole or hypersensitiveness to any drug
11. Patients who discontinued long-acting antipsychotics less than one treatment cycle before screening
12. Refractory schizophrenia patients who did not respond to treatments of two different type antipsychotics with adequate dose and course, or patients who did not respond to Clozapine
13. Patients who had Electroconvulsive Therapy (ECT) in the past 6 months After washout

1. Diagnosis of other mental diseases besides schizophrenia during the washout period 2. Significant abnormal ECG or laboratory examination results (ALT,AST>1.5 times of higher limit of normal range), not suitable to be enrolled based on the investigator's discretion.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-02; Study Completion 2005-07

PRIMARY OUTCOMES:
Deduction rate of PANSS total

SECONDARY OUTCOMES:
PANSS positive
PANSS negative
CGI
CGI improvement

CONTACTS AND LOCATIONS:
Overall Officials: Liang Shu, Professor, Principal Investigator — Institute of Mental Health, Peking University
Locations (6):
- China (6):
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - Psychiatry Dept. People's Hospital, Wuhan University, Wuhan, Hubei
  - Mental Health Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Anding Hosp. Capital University of Medical Science, Beijing
  - Institute of Mental Health, Peking University, Beijing
  - Shanghai Mental Health Center, Shanghai